CLINICAL TRIAL: NCT00842231
Title: Assessment of Visual Performance in Patients With Low Levels of Astigmatism
Status: Completed | Type: Observational
Sponsor: Alcon Research (Industry)
Responsible Party: Diane Houtman, OD, Associate Director, Surgical IOL Clinical Science, Alcon Research Ltd
Other Study IDs: P-08-06
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Results first posted 2010-09-08 (Estimated); Last update posted 2010-09-28 (Estimated); Status verified 2010-09

CONDITIONS: Cataract Extraction; Corneal Astigmatism
Keywords: Corneal astigmatism; post-cataract surgery; visual performance; Corneal astigmatism 0.5-0.75 Diopter
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Visual performance measures: Collection of visual performance measures in subjects with low levels of astigmatism.
  Interventions: Other: Visual performance measures

INTERVENTIONS:
Other: Visual performance measures — Collection of visual performance measures in subjects with low levels of astigmatism.

SUMMARY:
To assess visual performance in patients with low levels (0.5-0.75 Diopters) of corneal astigmatism.

ELIGIBILITY:
Inclusion Criteria:

* 50-75 years of age
* Proof of eye exam within the last 12 months
* Operated for uncomplicated, age-related cataracts >3 months
* Corneal astigmatism of 0.5-0.75 diopter

Exclusion Criteria:

* Previous ocular or refractive surgery/trauma
* Clinically severe corneal dystrophy
* Amblyopia
* Degenerative visual disorders

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects were selected from a single investigator's primary care clinic.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2009-01; Primary Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center For Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Visual Performance Measures
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Visual Performance Measures
Number analyzed (Participants) | 40
Age, Customized [Number; unit: Participants] — All patients were within the study inclusion/exclusion criteria and were within the ages of 50 and 75. No other specific age data is available.
  Participants | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: High and Low Contrast Acuity
Description: Visual acuity differences between subjects tested with full correction and spherical equivalent (SE) correction at contrast levels of 9% and 25% (low contrast acuity) and 100% (high contrast acuity). LogMAR is the "logarithm of the minimum angle of resolution". A lower logMAR value indicates better VA. These measurements were performed under photopic conditions by means of 9%, 25%, and 100% contrast ETDRS (Early Treatment Diabetic Retinopathy Study) charts (Vector Vision).
Time Frame: Day of study visit
Population: Data was collected for 40 eyes in 40 subjects. Only one operative eye of each subject was included in the study. If both eyes qualified, the dominant eye was selected.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Visual Performance Measures
Number analyzed (Participants) | 40
logMAR
  9% Contrast Acuity | 0.0855 (0.1111)
  25% Contrast Acuity | 0.065 (0.1019)
  100% Contrast Acuity | 0.082 (0.1013)

2. Primary Outcome: Contrast Sensitivity
Description: Contrast Sensitivity (CS) differences between subjects tested with full correction & spherical equivalent (SE) correction. CS is the measurement of one's ability to detect slight changes in luminance before it becomes indistinguishable. CS is measured in logarithmic units by means of an illuminated box, the CSV 1000 by Vector Vision. Testing was performed under photopic conditions (no glare) & mesopic conditions (with & without glare), and was measured at four spatial frequencies of 3, 6, 9, and 12 cycles per degree (cpd). A higher value for the logarithmic units translates to better CS.
Time Frame: Day of Study Visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Logrithmic Units
Arm/Group | Visual Performance Measures
Number analyzed (Participants) | 40
Logrithmic Units
  Mesopic 3 cycles per degree (cpd) | -0.047 (0.2917)
  Mesopic 6 cpd | 0.0896 (0.3575)
  Mesopic 9 cpd | 0.0038 (0.3597)
  Mesopic 12 cpd | -0.009 (0.371)
  Mesopic with glare 3 cpd | 0.0176 (0.2271)
  Mesopic with glare 6 cpd | 0.0241 (0.3146)
  Mesopic with glare 9 cpd | 0.0183 (0.2728)
  Mesopic with glare 12 cpd | 0.0669 (0.2559)
  Photopic 3 cpd | 0.0163 (0.2257)
  Photopic 6 cpd | 0.0181 (0.2539)
  Photopic 9 cpd | 0.0479 (0.3866)
  Photopic 12 cpd | 0.0321 (0.3215)

3. Primary Outcome: Reading Acuity and Speed
Description: Reading Acuity and Speed differences between subjects tested with full correction and spherical equivalent (SE) correction. Reading Acuity was measured using the Radner reading charts, which are logarithmically scaled at different acuity levels (print sizes), and expressed in terms of logRAD (logrithmic Reading Acuity Determination). Reading speed was measured in words per minute (wpm). The results were presented as Average Reading Speed by Print Size (logRAD).
Time Frame: Day of Study Visit
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: words per minute
Arm/Group | Visual Performance Measures
Number analyzed (Participants) | 40
words per minute
  logRAD Line -0.1 | 2.7469 [-33.4577 to 38.9515]
  logRAD Line 0 | 7.3292 [-10.7731 to 25.4315]
  logRAD Line 0.1 | 11.7498 [-0.7918 to 24.2914]
  logRAD Line 0.2 | 17.5404 [6.6243 to 28.4565]
  logRAD Line 0.3 | 10.1643 [-0.4353 to 20.7639]
  logRAD Line 0.4 | 13.4166 [3.2440 to 23.5892]
  logRAD Line 0.5 | 12.7487 [2.5761 to 22.9213]
  logRAD Line 0.6 | 11.9005 [1.8592 to 21.9419]
  logRAD Line 0.7 | 15.1714 [5.1301 to 25.2127]
  logRAD Line 0.8 | 9.7203 [-0.4523 to 19.8929]
  logRAD Line 0.9 | 11.4863 [1.3137 to 21.6589]
  logRAD Line 1.1 | 16.4043 [6.2317 to 26.5769]
  logRAD Line 1.2 | 8.8952 [-1.2774 to 19.0679]

ADVERSE EVENTS:
Description: This study consisted of a single visit on a single day. No adverse event data were collected.
Arm/Group | Visual Performance Measures
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No paper that incorporates Sponsor confidential information will be submitted for publication without Sponsor's prior written agreement.